CLINICAL TRIAL: NCT07255742
Title: Role of Lactoferrin in Prevention of Ventilator Associated Pneumonia in Neonates.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dalia Mohamed Salah (Other)
Responsible Party: Sponsor-Investigator, Dalia Mohamed Salah, Lecturer, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 36264PR702/5/24
Record Dates: First submitted 2025-11-16; First posted 2025-12-01 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-11

CONDITIONS: Ventilator Associated Pneumonia
Keywords: Lactoferrin,VAP
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Lactoferrin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lactoferrin group (Experimental): Neonates who will receive oral lactoferrin supplementation.
  Interventions: Dietary Supplement: Lactoferrin in prevention of VAP
- Control (Other): who Will not receive
  Interventions: Other: Control

INTERVENTIONS:
Dietary Supplement: Lactoferrin in prevention of VAP — oral dose separate from feeds [at a daily dose of 100mg/day] via orogastric tube from first day of enrollment till time of successful extubation plus standard preventive measures of VAP; these include semi recumbent position, hand washing, suctioning when needed, endotracheal tube with subglottic secretion drainage, using heat and moisture exchanger filter, oral hygiene, changing of tubes only when needed and changing of ventilator circuit every 5 days.
  Arms: Lactoferrin group
Other: Control — They will receive standard preventive VAP strategies only.
  Arms: Control

SUMMARY:
The aim of the study is to

1. Evaluate the preventive value of Lactoferrin on VAP among ventilated neonates.
2. Evaluate the Primary outcome of Lactoferrin on:

   Sepsis, Feeding intolerance, Vomiting, Constipation or diarrhea
3. Evaluate the effect of Lactoferrin in critically ventilated neonates on:

Incidence of VAP Duration of mechanical ventilation Duration of hospital stay

DETAILED DESCRIPTION:
Randomised controlled trial

ELIGIBILITY:
Inclusion Criteria:

Preterm neonates requiring mechanical ventilation.

Gestational age: (GA 28-36 weeks).

Expected need for mechanical ventilation for ≥ (48hours)

Exclusion Criteria:

Congenital anomalies of the lung or airway.

Major congenital heart disease.

Proven early-onset sepsis at enrollment.

Severe perinatal asphyxia (e.g., Apgar < 3 at 5 minutes or seizures).

Known contraindication or allergy to lactoferrin.

Severe gastrointestinal pathology (e.g., NEC stage II or higher).

Any condition deemed by the clinical team to interfere with study participation.

Ages: 0 Days to 90 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-04 (Actual)

PRIMARY OUTCOMES:
Prevention of VAP | From enrollment until day 28 of life or NICU discharge, whichever occurs first.
  Diagnosis of VAP using the CDC/NHSN clinical and radiological criteria for neonatal ventilator-associated events. Outcome measured as the percentage (%) of enrolled neonates who develop VAP during NICU stay or up to 28 days of life.
Prevention of VAP | during NICU stay
  Incidence of ventilator-associated pneumonia during mechanical ventilation.

CONTACTS AND LOCATIONS:
Locations (1):
- Neonatal Intensive Care Unit, Tanta University Children's Hospital, Tanta, Egypt